CLINICAL TRIAL: NCT06662708
Title: Accurate Prediction and Treatment of Prostate Cancer by Artificial Intelligence Model-based Whole Slide Images and MRIs
Brief Title: Artificial Intelligence Models for Precision Prediction and Treatment of Prostate Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shao Pengfei (Other)
Collaborators: Institute of Automation, Chinese Academy of Sciences (Other)
Responsible Party: Sponsor-Investigator, Shao Pengfei, Chief physician, The First Affiliated Hospital with Nanjing Medical University
Organization: The First Affiliated Hospital with Nanjing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: Shao Pengfei
Record Dates: First submitted 2024-08-13; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Prostate Cancer; Prostate Intraductal Carcinoma; Prostate Cancer Aggressiveness; Prostate Cancer Stage; Pathology
Keywords: Articicial Intelligence; Whole Slide Image; mp-MRI; Prostate Cancer; Prediction Model
MeSH Terms: conditions — Prostatic Neoplasms; Prostate Cancer, Hereditary, 7

STUDY DESIGN:
Intervention Model Description: Inclusion of enrolled patients in an artificial intelligence predictive model that predicts postoperative pathology, precise preoperative diagnosis (including benign and malignant, invasive, grading, and subtypes) or 3D lesion modelling based on the information provided
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): This group of patients will receive predictions assisted by artificial intelligence models.
  Interventions: Diagnostic Test: Accurate Prediction Artificial Intelligence Models
- Control Group (No Intervention): This group of patients will not receive predictions assisted by artificial intelligence models.

INTERVENTIONS:
Diagnostic Test: Accurate Prediction Artificial Intelligence Models — Diagnostic Test: Accurate Prediction Artificial Intelligence Models Post-operative pathology, precise pre-operative diagnosis (including benign and malignant, invasive, grading, subtypes) or 3D lesion modelling will be predicted based on the AI predictive model in response to the information provided
  Arms: Experimental group

SUMMARY:
The aim of this clinical trial is whether artificial intelligence models can be used for accurate clinical preoperative diagnosis and postoperative diagnosis of pathological findings, and will also measure the accuracy of the predictions made by the artificial intelligence models.The main target questions addressed by the model building are:

1. whether the AI model can learn from preoperative MRI and postoperative Whole Slide Images so as to accurately predict information such as benignness or malignancy, aggressiveness, grading, subtypes, genes, etc. for participants suspected of having prostate cancer preoperatively/puncturally.
2. whether the AI model is capable of learning postoperative macropathology slides to enable outcome diagnosis of surgical pathology slides in new participants.

Participants will:

1. complete an MRI examination and have their MRI images analysed by the established AI model to make an accurate diagnosis of them.
2. Based on the diagnosis, if prostate cancer is predicted, they will undergo radical prostate cancer surgery and refine their surgical pathology.

DETAILED DESCRIPTION:
Based on artificial intelligence technology, the prediction model is built by outlining the quantitative mapping correlation between annotated prostate cancer Whole Slide Images and MRI, and clarifying the common features. Firstly, the model can accurately diagnose the radical pathology of prostate cancer, which can be exempted from immunohistochemistry to obtain detailed pathological information; secondly, the established AI prediction model can accurately diagnose the benign/malignant, invasiveness, grade and subtype of prostate cancer by predicting the participant's MRI images before surgery or puncture, so that a personalised treatment plan can be formulated for the patient before operation or puncture. Finally, based on AI technology, the model learns from the MRI images and performs 3D reconstruction of the prostate and lesions before surgery/puncture, thus clarifying the exact location of the lesions and guiding puncture or surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected PCa (elevated PSA or suspicious positive lesions on ultrasound or MRI results);

Exclusion Criteria:

* Previous treatment of the prostate in any form, including surgery, radiotherapy/chemotherapy, endocrine therapy, targeted therapy and immunotherapy;
* Patients with any item missing from the baseline clinical and pathological information;
* Patients with a history of other malignancies, serious comorbidities or other health problems;
* Unable to provide/sign an informed consent form;
* Patients who, in the judgement of the investigator, are deemed unfit to participate in this clinical trial;

Min Age: 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Prediction of postradical prostate cancer pathology after radical prostatectomy using the 'AUC' comprehensive assessment model | From subject enrolment to initial post-surgery, usually 30-90 days.
  'AUC' refers to the area under the ROC (Receiver Operating Characteristic) curve, which indicates the performance of the model in predicting immunohistochemistry-related pathological information of prostate cancer after surgery, and the AUC ranges from 0-1, with the larger value indicating the better prediction effect.
Predicting the performance of post-radical pathology by the 'AUC' comprehensive assessment model | From subject enrolment to initial post-surgery, usually 30-90 days.
  'AUC' refers to the area under the ROC (Receiver Operating Characteristic) curve, indicating the level of performance of the model in predicting prostate cancer in the preoperative period, with AUC ranging from 0-1, with larger values indicating better prediction results.
'F1 Score' to assess performance of preoperative 3D modelling | From subject enrolment to initial post-surgery/puncture recovery, usually 30-90 days.
  A reconciled average of the preoperative 3D modelling precision and recall assessed through the 'F1 score', which represents the match to the real situation.

SECONDARY OUTCOMES:
Assess the amount of cost difference between the predictive model and the clinical approach by "economic cost savings" | From subject enrolment to initial post-surgery/puncture recovery, usually 30-90 days.
  Compare the difference in costs incurred using a predictive model with those predicted using a clinical approach, the difference will be in yuan.
"Diagnostic Time" evaluate the time taken to predict immunohistochemistry-related pathology in the postoperative period. | From subject enrolment to initial post-surgery/puncture recovery, usually 30-90 days.
  The time spent postoperatively predicting or assisting the pathologist in obtaining immunohistochemistry-related pathology information is assessed by "Diagnostic Time" and will be measured in minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University (Jiangsu Provincial People's Hospital), Nanjing, Jiangsu, China